CLINICAL TRIAL: NCT04456517
Title: REACT Trial: A Randomized, Double Blind, Placebo-controlled, Crossover Study of Ranolazine for the Treatment of Crohn's Disease-associated Diarrhea
Brief Title: Reduce Crohn's-Associated Diarrhea With Sodium Channel Therapy
Acronym: REACT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual and subject engagement
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Dawn Beaulieu, Principle Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200640
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Crohn's Disease; Inflammatory Bowel Disease
Keywords: Diarrhea
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Diarrhea | interventions — Ranolazine

STUDY DESIGN:
Intervention Model Description: Participants receive one of two alternative interventions during the initial phase of the study and receive the other intervention during the second phase of the study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ranolazine, Then Placebo (Experimental): - Participants first receive a Ranolazine 500 mg tablet twice daily for 12 weeks, they then receive a Placebo tablet (matching Ranolazine 500 mg tablets) twice daily for 12 weeks. This treatment will be given to participants with either active CD or patients with CD that is in remission but who experience continued symptoms
  Interventions: Drug: Ranolazine; Drug: Placebo
- Placebo, Then Ranolazine (Experimental): - Participants first receive a Placebo tablet (matching Ranolazine 500 mg tablets) twice daily for 12 weeks, they then receive a Ranolazine 500mg tablet twice daily for 12 weeks. This treatment will be given to participants with either active CD or patients with CD that is in remission but who experience continued symptoms
  Interventions: Drug: Ranolazine; Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — 500 mg tablet
Drug: Placebo — Ranolazine-matched placebo tablet

SUMMARY:
Crohn's disease is an inflammatory disorder that can affect any part of the gastrointestinal (GI) tract. Some patients still experience persistent diarrhea or other symptoms such as abdominal pain even when their Crohn's disease is in remission. Diarrhea and/or abdominal pain that is not responsive to standard therapies can significantly affect a patient's quality of life and ability to work. The purpose of this study is to test the safety and effectiveness of the drug ranolazine in reducing Crohn's disease-associated diarrhea and other symptoms. Ranolazine is approved by the US Food & Drug Administration (FDA) for chronic angina (a heart condition). This study is investigating if ranolazine could be used in the setting of Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Meet diagnostic criteria for Crohn's Disease with active diarrhea Either with active disease or in remission (as defined by endoscopic or radiographic findings) but experiencing symptoms (e.g., diarrhea, abdominal pain)
* Have greater than three loose stools per day

Exclusion Criteria:

* Male and female subjects <18 years of age
* Significant change in medication including prednisone, antidepressant medications, or stimulants within the last 4 weeks

  a. Allowances include: Rectal hydrocortisone, rectal mesalamine, addition of prednisone (up to 20mg) for flares, etc.
* Regular (daily) use of opioids or other drugs of abuse including heavy alcohol or marijuana use
* Severe psychiatric disease including schizophrenia, psychosis, suicidal depression
* Previous use of ranolazine within 2 months prior to enrollment
* Prior use of ranolazine which was discontinued for safety or tolerability
* Metabolic derangement defined as liver function tests >3x upper limit of normal or severe renal disease defined as calculated creatinine clearance <30 mL/min
* Have liver cirrhosis
* Concurrent use of CYP3A inhibitors, inducers, or substrates

  a. These may include: ketoconazole, itraconazole, nefazodone, nelfinavir, ritonavir, indinavir, and saquinavir, clarithromycin, or rifampin, rifapentine, phenobarbital, phenytoin, and St. John's Wort, digoxin.
* A family history of (or congenital) long QT syndrome or known acquired QT interval prolongation
* Inability or refusal to give informed consent for any reason including a diagnosis of dementia or cognitive impairment
* Patients who are pregnant or breastfeeding
* Patients who are enrolled in other investigational drug studies or who have taken investigational drugs within 30 days before enrollment
* Other factors which in the opinion of the investigator could potentially impact the study outcomes (e.g., underlying disease, medications, history) or prevent the participant from completing the protocol (poor compliance or unpredictable schedule)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn B. Beaulieu, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators agree to the timely release and sharing of information to be no later than the acceptance for publication of the main findings from the final data set. Investigators are also committed to ensuring that all data are free of identifiers that would permit linkage to individual research participation as well as variables that could lead to deductive disclosure of individual subjects.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 of 4 participants were randomized.
Period: First Intervention:Baseline to 12 Weeks
Arm/Group | Ranolazine, Then Placebo | Placebo, Then Ranolazine
Started | 3 | 1
Completed | 3 | 0
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Second Intervention: 12 Weeks to 24 Week
Arm/Group | Ranolazine, Then Placebo | Placebo, Then Ranolazine
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranolazine, Then Placebo | Placebo, Then Ranolazine | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (9.5) | 59 (9.1) | 43 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 1 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Daily Number of Loose Stools
Description: Daily number of loose stools will be collected directly from all subjects using MyCap.
Time Frame: Baseline to 12 weeks
Population: 1 subject in Placebo arm only has baseline data since they withdrew.
Measure: Mean (Standard Deviation); unit: number of liquid stools
Groups:
- Ranolazine: - Participants receive a Ranolazine 500 mg tablet twice daily for 12 weeks.
- Placebo: - Participants receive a Placebo tablet (matching Ranolazine 500 mg tablets) twice daily for 12 weeks.
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 3 | 4
number of liquid stools
  Liquid Stools at Baseline | 3.6 (2.5) | 4.5 (3.4)
  Liquid stools at Week 12: number analyzed (Participants) | 3 | 3
  Liquid stools at Week 12 | 2.9 (1.6) | 3.2 (0.8)

2. Secondary Outcome: Crohn's Disease Activity Index (CDAI) Score
Description: The Crohn's Disease Activity Index (CDAI) combines weighted scores of clinical and laboratory variables to estimate disease severity. The CDAI consists of eight variables, two of which are subjective, related to the disease, each weighted according to its ability to be predictive of disease activity. The absolute score ranges from 0 to 600. CDAI scores of less than 150 indicate a clinical remission and scores over 450 indicate severely active disease. Since blood draws will not be performed as part of this study, the hematocrit component of the CDAI will not be assessed.
Time Frame: Baseline to 12 weeks
Population: One of three subjects on ranolazine did not have a baseline CDAI score. 1 of 4 subject on placebo did not complete course.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Ranolazine: - Participants first receive a Ranolazine 500 mg tablet twice daily for 12 weeks.
- Placebo: - Participants first receive a Placebo tablet (matching Ranolazine 500 mg tablets) twice daily for 12 weeks.
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 3 | 4
score on a scale
  Baseline CDAI: number analyzed (Participants) | 2 | 4
  Baseline CDAI | 169 (90.5) | 117 (88.1)
  12 week CDAI: number analyzed (Participants) | 3 | 3
  12 week CDAI | 100 (99.6) | 110.3 (97.8)

3. Secondary Outcome: Harvey Bradshaw Index (HBI) Score
Description: The Harvey-Bradshaw index (Harvey-Bradshaw Index - HBI) assesses the degree of illness (activity) in patients with Crohn's disease. The HBI consists of 5 items with a minimum score of 0 and a maximum attainable score depending on the number of stools the patient identifies per day. HBI scores < 5 are defined as clinical remission, HBI between 5 and 7 as mild disease, HBI between 8 and 16 as moderate disease, and HBI > 16 as severe disease.
Time Frame: Baseline to Week 12
Population: 1 of 4 subjects assigned placebo for 12 weeks did not complete course.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 3 | 4
score on a scale
  Baseline HBI | 6.7 (1.5) | 5 (3.1)
  12 week HBI: number analyzed (Participants) | 3 | 3
  12 week HBI | 4.7 (3.5) | 5 (1.7)

4. Secondary Outcome: Short Inflammatory Bowel Disease Questionnaire (SIBDQ) Score
Description: The SIBDQ is a 10-item questionnaire measuring quality of life in four domains: bowel symptoms, emotional health, systemic symptoms, and social function and is scored on a 7-point Likert scale from 1 (severe problem) to 7 (no problems at all). The absolute score ranges are from 10 (poor Health-related quality of life) to 70 (optimum Health-related quality of life).
Time Frame: Baseline to 12 weeks
Population: 1 of 4 subjects in placebo arm did not complete course.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 3 | 4
score on a scale
  Baseline SIBDQ | 52 (10.5) | 54 (10.1)
  Week 12 SIBDQ: number analyzed (Participants) | 3 | 3
  Week 12 SIBDQ | 57.3 (8.1) | 59.3 (5.9)

5. Secondary Outcome: Patient Health Questionnaire (PHQ-9) Score
Description: The PHQ-9 is a 9-item questionnaire that screens for the presence and severity of depression and can be used to make a depression diagnosis using DSM-IV criteria.
  The PHQ-9 is scored on a 3-point Likert scale from 0 (not at all) to 3 (nearly every day). The absolute score ranges are from 0 (none or minimal depression) to 27 (severe depression).
Time Frame: Baseline to week 12
Population: 1 of 4 subjects in placebo arm did not complete course.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 3 | 4
score on a scale
  Baseline PHQ9 | 8.3 (5.5) | 7 (3.9)
  12 week PHQ9: number analyzed (Participants) | 3 | 3
  12 week PHQ9 | 5.7 (3.5) | 6.3 (3.8)

ADVERSE EVENTS:
Time Frame: Baseline to 24 weeks
Description: Adverse event information was collected for any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Groups:
- Placebo: Participants receive a Placebo tablet (matching Ranolazine 500 mg tablets) twice daily for 12 weeks.
Arm/Group | Ranolazine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine (N=3) | Placebo (N=4)
Blurry vision (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT04456517/Prot_SAP_001.pdf
  • Informed Consent Form (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/17/NCT04456517/ICF_002.pdf